CLINICAL TRIAL: NCT05724511
Title: Department of Nutrition, China Medical University
Brief Title: The Effect of Probiotics on Depression Syndrome and Risk Factors of Cardiovascular Disease in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Pei-Yu Wu, Project Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMUH111-REC3-178
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Depression Mild; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: MIYAIRI 588
- Control (No Intervention)

INTERVENTIONS:
Drug: MIYAIRI 588 — In the 3 months intervention, each subjects take 1g/package with meal, and 3 packages/day.
  Arms: Intervention

SUMMARY:
As the investigators know, only few researches focus on the effect of probiotics on depression in hemodialysis patients. Besides, probiotics also have benefit effect on dyslipidemia and hypertension in general population. Both of them are the risk factors of cardiovascular disease which is the major cause of death in hemodialysis patients. Therefore, this study looks for the effect of probiotics on depression syndrome and risk factors of cardiovascular disease in hemodialysis patients. This is a randomized controlled trial. All patients will be assigned at random to intervention group or control group. This study plans to recruit 70 hemodialysis patients and expects at least 30 patients in each group at the end of study period. The investigators provide probiotics (C. butyricum MIYAIRI 588) to intervention group and provide nothing to the control group.

All patients need to maintain the lifestyle during study period. Genomic analysis of gut microbiota on patients' fecal samples will be used to evaluation their compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older undergoing hemodialysis (at least 3 months), 3 times per week, and URR ≥65%

Exclusion Criteria:

1. allergic to the components of the intervention drug, low tolerance of milk or dairy products
2. Has the diagnosis of dementia, delirium, bipolar disorder, schizophrenia, or liver failure
3. Beck Depression Inventory Chinese version 2.0 score higher than 14, or has significant suicide risk during study
4. Following significantly clinical syndrome: obsessive compulsive disorder, schizoid personality disorder, schizotypal personality, paranoid、antisocial Personality Disorder, histrionic personality disorder
5. With addiction to alcohol or drugs, terminal cancer, severe infection, heart failure, central venous catheter in the past 6 months
6. Taking antibiotics, anti-oxidant vitamin supplement, probiotics, prebiotics, antidepressants, anti-anxiety medicine, yogurt and the products in the past 3 months
7. Pregnant or lactating

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The change of depression score | Change from Baseline depression score at 3 months
  Beck Depression Inventory score (Chinese version 2.0). The score range is from 0 to 63, and the higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
We have promised our subjects that all of their information will be protected, and this is included in the Informed Consent Form.